CLINICAL TRIAL: NCT05504226
Title: A Multicenter, Randomized, Placebo-controlled, Parallel Group, Double-blind, Phase III Study to Evaluate the Efficacy and Safety of Teneligliptin in Patients With Type 2 Diabetes Who Have Inadequate Glycemic Control With Metformin and Empagliflozin 25 mg
Brief Title: Clinical Efficacy and Safety Evaluation of Teneligliptin in Type 2 Diabetes Who Have Inadequate GlycemIc Control With Empaglyflozin 25 mg and Metformin
Acronym: TERA 305
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HD-MP-305
Record Dates: First submitted 2022-08-11; First posted 2022-08-17 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teneligliptin 20 mg (Experimental)
  Interventions: Drug: Teneligliptin (as Teneligliptin Hydrobromide) 20 Mg Oral Tablet
- Teneligliptin placebo (Placebo Comparator)
  Interventions: Drug: Teneligliptin Placebo Oral Tablet

INTERVENTIONS:
Drug: Teneligliptin (as Teneligliptin Hydrobromide) 20 Mg Oral Tablet — To be orally administered once daily for 52 weeks.
  Arms: Teneligliptin 20 mg
Drug: Teneligliptin Placebo Oral Tablet — To be orally administered once daily for 52 weeks. This arm will be switched to teneligliptin from week 24.
  Arms: Teneligliptin placebo

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of teneligliptin 20 mg orally administered once daily for 24 weeks compared with placebo in patients with type 2 diabetes mellitus who have inadequate glycemic control with empaglyflozin 25 mg and metformin

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type II diabetes mellitus aged 19 years or older
* Subjects with 7.0%≤HbA1c≤10.5% at screening visit
* Subjects with fasting plasma glucose ≤ 270mg/dL at screening visit

Exclusion Criteria:

* Subjects with type 1 diabetes mellitus or secondary diabetes
* Subjects with history of diabetic ketoacidosis, diabetic coma or pre-coma, lactic acidosis, and acute or chronic acidosis within 6 months prior to the screening visit
* Subjects who have been administered with weight-loss drug (e.g., orlistat, phentermine/topiramate, lorcaserin)
* Body mass index greater than 40 kg/m2 at the screening visit
* Subjects with heart failure (Class III-IV of NYHA classification) or arrhythmia that requires treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Changes from baseline HbA1c at week 24 | Baseline (week 0) and week 24

SECONDARY OUTCOMES:
Changes from baseline FPG at week 24 | Baseline (week 0) and week 24
Percentage of subjects achieving the HbA1c goals (HbA1c < 7.0% or < 6.5%) at week 24 | Baseline (week 0) and week 24
Changes from baseline in BMI at week 24 | Baseline (week 0) and week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided